CLINICAL TRIAL: NCT04986423
Title: A Randomized Phase 2b Study of ZEN003694 in Combination With Enzalutamide Versus Enzalutamide Monotherapy in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: ZEN003694 and Enzalutamide Versus Enzalutamide Monotherapy in Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zenith Epigenetics (Industry)
Collaborators: Astellas Pharma Inc (Industry); Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEN003694-201
Record Dates: First submitted 2021-07-14; First posted 2021-08-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: mCRPC; ZEN003694; ZEN-3694; Bromodomain; BETi; Enzalutamide; Xtandi®
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A - ZEN003694 + Enzalutamide (Experimental): Patients will be administered enzalutamide (160 mg) orally once daily for 21 days prior to the initiation of the combination therapy (Lead-in) to reach steady state concentration (Css) prior to Cycle 1. After the Lead-in, ZEN003694 (72 mg) will be administered orally one daily in combination with daily enzalutamide for 28-day cycles.
  Interventions: Drug: ZEN003694; Drug: Enzalutamide
- Cohort A - Enzalutamide (Active Comparator): Patients will be administered enzalutamide (160 mg) orally once daily for 21 days prior to Cycle 1 Day 1 (Lead-in). After the Lead-in, patients will be administered enzalutamide 160 mg orally once daily for 28-day cycles. Active control patients will have the option to cross-over to treatment with ZEN003694 in combination with enzalutamide upon confirmed radiographic progression by PCWG3 criteria by independent central review.
  Interventions: Drug: Enzalutamide
- Cohort B - ZEN003694 + Enzalutamide (Experimental): Patients will be administered enzalutamide (160 mg) orally once daily for 21 days prior to the initiation of the combination therapy (Lead-in) to reach steady state concentration (Css) prior to Cycle 1. After the Lead-in, ZEN003694 (72 mg) will be administered orally one daily in combination with daily enzalutamide for 28-day cycles.
  Interventions: Drug: ZEN003694; Drug: Enzalutamide
- Cohort B - Enzalutamide (Active Comparator): Patients will be administered enzalutamide (160 mg) orally once daily for 21 days prior to Cycle 1 Day 1 (Lead-in). After the Lead-in, patients will be administered enzalutamide 160 mg orally once daily for 28-day cycles. Active control patients will have the option to cross-over to treatment with ZEN003694 in combination with enzalutamide upon confirmed radiographic progression by PCWG3 criteria by independent central review.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: ZEN003694 — 72 mg PO QD
  Other Names: ZEN-3694
  Arms: Cohort A - ZEN003694 + Enzalutamide; Cohort B - ZEN003694 + Enzalutamide
Drug: Enzalutamide — 160 mg PO QD
  Other Names: Xtandi®; MDV3100

SUMMARY:
This is an open-label, randomized, Phase 2b study of ZEN003694 in combination with enzalutamide vs. enzalutamide monotherapy in patients with mCRPC who have progressed on prior abiraterone by PCWG3 criteria. Disease must have progressed on only abiraterone by PCWG3 criteria prior to study entry.

The patient population will be separated into two cohorts:

Cohort A: Patients with poor response to prior abiraterone defined as:

* Abiraterone started in hormone-sensitive prostate cancer (HSPC) disease setting: < 12 months duration on abiraterone or failure to achieve PSA nadir of 0.2 ng/mL while taking abiraterone, or;
* Abiraterone started in castrate-resistant prostate cancer (CRPC) disease setting: < 6 months duration on abiraterone or failure to achieve PSA50 response while on abiraterone

Cohort B: Patients with response to prior abiraterone, defined as:

* Abiraterone started in hormone-sensitive prostate cancer (HSPC) disease setting: ≥ 12 months duration on abiraterone and nadir PSA < 0.2 ng/mL, or;
* Abiraterone started in castrate-resistant prostate cancer (CRPC) disease setting: ≥ 6 months duration on abiraterone and confirmed PSA50 response

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 years
2. Metastatic, castration-resistant, histologically confirmed prostate cancer
3. Surgical castration or continuous medical castration for ≥ 8 weeks prior to screening; serum testosterone < 50 ng/dL confirmed within 4 weeks of first administration of study drug
4. Have progressed on prior abiraterone treatment by PCWG3 criteria
5. Patients who are not candidates for chemotherapy in the opinion of the investigator or patients who decline chemotherapy
6. Cohort A only - Patient must meet definition of poor responder to abiraterone by one of the following:

   1. Abiraterone started in hormone-sensitive prostate cancer (HSPC) disease setting: < 12 months duration on abiraterone or failure to achieve PSA nadir of 0.2 ng/mL while taking abiraterone
   2. Abiraterone started in castrate-resistant prostate cancer (CRPC) disease setting: < 6 months duration on abiraterone or failure to achieve a PSA50 response
7. Cohort B only - Patient must meet definition of responder to abiraterone by one of the following:

   1. Abiraterone started in hormone-sensitive prostate cancer (HSPC) disease setting: ≥ 12 months duration on abiraterone and nadir PSA < 0.2 ng/mL
   2. Abiraterone started in castrate-resistant prostate cancer (CRPC) disease setting: ≥ 6 months duration on abiraterone and PSA50 response
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

1. Any history of brain metastases, prior seizure, conditions predisposing to seizure activity
2. Have previously received an investigational BET inhibitor (including previous participation in this study or a study of ZEN003694)
3. Receipt of prior second-generation androgen receptor inhibitors (e.g. enzalutamide, apalutamide, darolutamide, proxalutamide). Receipt of first-generation AR antagonists (e.g. bicalutamide, nilutamide, flutamide) does not count towards this limit.
4. Have received prior chemotherapy in the metastatic castration-resistant setting (prior chemotherapy in the hormone-sensitive setting is allowed provided last dose was at least 6 months prior to first dose of study drug)
5. Have received prior systemic anti-cancer therapy within 2 weeks or five half-lives, whichever is shorter, prior to the first administration of study drug
6. Have received exogenous administration of testosterone therapy since discontinuation of abiraterone.
7. Failure to recover to Grade 1 or lower toxicity related to prior systemic therapy (excluding alopecia and neuropathy) prior to study entry
8. Radiation therapy within 2 weeks of the first administration of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Radiographic progression-free survival (rPFS) by BICR | Randomization up to 30 months
  Time from date of randomization to the date of first disease radiographic progression or death for any reason. Radiographic progression disease will be evaluated by RECIST 1.1 and PCWG3.

SECONDARY OUTCOMES:
Cohorts A + B: Radiographic progression-free survival (rPFS) by BICR | Randomization up to 30 months
  Time from date of randomization to the date of first disease radiographic progression or death for any reason. Radiographic progression disease will be evaluated by RECIST 1.1 and PCWG3
Cohort A: Radiographic progression-free survival (rPFS) by investigator assessment | Randomization up to 30 months
  Time from date of randomization to the date of first disease radiographic progression or death for any reason. Radiographic progression disease will be evaluated by RECIST 1.1 and PCWG3.
Cohort A + B: Radiographic progression-free survival (rPFS) by investigator assessment | Randomization up to 30 months
  Time from date of randomization to the date of first disease radiographic progression or death for any reason. Radiographic progression disease will be evaluated by RECIST 1.1 and PCWG3.
Cohort A: Progression-free survival (PFS) by investigator assessment | Randomization up to 30 months
  Time from date of randomization to the date of first disease radiographic progression, clinical progression, or death for any reason. Radiographic progression of disease will be evaluated by RECIST 1.1 and PCWG3 by investigator assessment. Clinical progression is significant pain increase or clinical deterioration that requires initiating another line of treatment.
Cohort A + B: Progression-free survival (PFS) by investigator assessment | Randomization up to 30 months
  Time from date of randomization to the date of first disease radiographic progression, clinical progression, or death for any reason. Radiographic progression of disease will be evaluated by RECIST 1.1 and PCWG3 by investigator assessment. Clinical progression is significant pain increase or clinical deterioration that requires initiating another line of treatment.
Cohort A: Overall survival (OS) | Randomization up to 30 months
  Time from date of randomization to the date of death from any cause
Cohort A + B: Overall survival (OS) | Randomization up to 30 months
  Time from date of randomization to the date of death from any cause
Cohort A: PSA50 response rate | Randomization up to 30 months
  PSA response is a reduction in serum PSA concentration of ≥50% from baseline.
Cohort A + B: PSA50 response rate | Randomization up to 30 months
  PSA response is a reduction in serum PSA concentration of ≥50% from baseline.
Cohort A: Assess efficacy endpoints for patients enrolled in the USA | Randomization up to 30 months
Cohort A + B: Assess efficacy endpoints for patients enrolled in the USA | Randomization up to 30 months
Objective response rate (ORR) | Randomization up to 30 months
  Proportion of the patients who have either a complete response (CR) or partial response (PR) by RECIST 1.1 criteria who have measurable disease at baseline.
Patient-reported health status and quality of life (QoL) measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Screening and Day 1 of every 28-day Cycle up to 30 months
  EORTC QLQ-C30: cancer-specific instrument with 30 questions to assess the participant QoL. First 28 questions used to evaluate 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, nausea and vomiting, pain) and other single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Each question assessed on a 4-point scale (1= not at all, 2= a little, 3= quite a bit, 4= very much); functional scales: higher score = better level of functioning; symptom scale: higher score = more severe symptoms; for single items: higher score= more severe problem. Last 2 questions used to evaluate global health status (GHS)/QoL. Each question was assessed on 7-point scale (1= very poor to 7= excellent). Scores averaged, transformed to 0-100 scale; higher score=better quality of life/better level of functioning.
Patient-reported health status and quality of life (QoL) measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Prostate Module (EORTC QLQ-PR25). | Screening and Day 1 of every 28-day Cycle up to 30 months
  EORTC QLQ-PR25: prostate cancer specific instrument with 25 questions used in conjunction with EORTC QLQ-C30 to assess the participant QoL. Used to evaluate 5 multi-item scales (urinary, bowel, and hormonal treatment-related symptoms, sexual activity, and sexual functioning) and one single item (problems due to incontinence aid use). Each question assessed on a 4-point scale (1= not at all, 2= a little, 3= quite a bit, 4= very much). Scores averaged, transformed to 0-100 scale; higher score=better quality of life/better level of functioning.
Time to initiation of chemotherapy | Randomization up to 30 months
  Time from date of randomization to the first dose of chemotherapy.
Time to first skeletal related event (SRE) | Randomization up to 30 months
  Time from date of randomization to the first SRE such as pathological fracture, surgery/radiotherapy for pain/prevention of fracture, hypercalcemia, and spinal cord compression.
Measure plasma concentrations of ZEN003694 and the active metabolite ZEN003791 | Cycle 1 Day 1: Pre-dose, 1 hour, 2 hours, and 4 hours post-dose; Cycle 2 Day1: Pre-dose, 1 hour, 2 hours, and 4 hours post-dose
  Plasma concentrations of ZEN003694 and the active metabolite ZEN003791 will be measured.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (16):
  - California Research Institute, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Innovative Clinical Research Institute, Whittier, California
  - Colorado Urology, Lakewood, Colorado
  - D&H Cancer Research Center, LLC, Margate, Florida
  - BRCR Global, Plantation, Florida
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Urology Associates, P.C., Nashville, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- China (15):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotang University, Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No